CLINICAL TRIAL: NCT06640322
Title: Turkish Validity and Reliability of the Craniocervical Dysfunction Index in Patients With Non-specific Neck Pain
Brief Title: Craniocervical Dysfunction Index in Turkish Patients With Non-specific Neck Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayse Unal, Assoc. Prof., Alanya Alaaddin Keykubat University
Other Study IDs: 11.10.2024/CDI-NNP
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain; Craniocervical Disfunction
Keywords: Neck Pain; Craniocervical Disfunction; Reliability; Validity
MeSH Terms: conditions — Neck Pain | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reliability and validity — Reliability and validity of Craniocervical Dysfunction Index in Turkish Patients With Non-specific Neck Pain

SUMMARY:
The aims of this study were to perform cultural adaptation of the Craniocervical Dysfunction Index in patients with non-specific neck pain, reliability and validity of the index Turkish speaking adults.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-60 years
* Clinical diagnosis of non-specific neck pain
* Being able to communicate in Turkish
* Volunteering to participate in the study

Exclusion Criteria:

* Over 60 years of age
* Those with impairments in cervical mobility that affected the postural assessment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: aproximately 5o patients with non-specific neck pain between the ages of 20-60 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Craniocervical Dysfunction Index | Baseline
  The assessment of craniocervical dysfunction is performed objectively and comprehensively through the Craniocervical Dysfunction Index (CDI), which was developed based on the Helkimo Dysfunction Index. The CDI numerically grades the severity of the functional disorders of the cervical spine. Through this index it is possible to assess the craniocervical dysfunction, regardless of the opinion of the patients, of the severity of the symptoms, and of the need for treatment. The CDI objectively indicates the dysfunction of the cervical region by numerical average, assessing the degree of dysfunction and enabling the differential diagnosis, suggesting the priority and monitoring of the treatment these changes may be reassessed over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaadin Keykubat University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No